CLINICAL TRIAL: NCT01327274
Title: Phase 3 Multicenter Study of Magnetic Mini-Mover for Pectus Excavatum
Brief Title: Multicenter Trial of Magnetic Mini-Mover for Pectus Excavatum
Acronym: 3MP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Harrison (Other)
Collaborators: Shriners Hospitals for Children (Other); Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor-Investigator, Michael Harrison, Professor of Surgery and Pediatrics, Emeritus, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FD003341-03-06; FD-R-01FD-03341 (Other Grant/Funding Number: FDA)
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Pectus Excavatum
Keywords: Pectus excavatum; Chest wall deformity; Magnetic Mini-Mover Procedure; Pectus Severity Index; pediatric medical device; magnetic alteration; sunken chest
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): This is a non-randomized study in which otherwise healthy patients, ages 8-14, with severe pectus excavatum (PSI > 3.5) will undergo the interventional treatment arm by having outpatient surgery and the Magnetic MIni-Mover Magnimplant procedure is performed during which the magnetic implant is surgically placed. After 2 years of treatment with the implanted magnet and brace treatment, the Magnetic Mini-Mover Magnimplant will be explanted. After surgery and recovery, all subjects will be fitted for an orthotic brace, which houses the external magnet and records brace-wear compliance. They will undergo 3MP treatment for 18-24 months, enough to attempt to improve their PSI (< 3.25).
  Interventions: Device: Magnetic Mini-Mover Procedure (Magnimplant)

INTERVENTIONS:
Device: Magnetic Mini-Mover Procedure (Magnimplant) — This is a non-randomized study in which otherwise healthy patients, ages 8-14, with severe pectus excavatum (PSI > 3.5) will undergo the Magnetic Mini-Mover procedure outpatient surgery. The Magnimplant or Magnetic Mini-Mover device implant will surgically implanted on the sternum. Patients will be required to wear a custom-fitted orthotic brace, which houses the external magnet and records brace-wear compliance. They will undergo brace treatment for 18-24 months, enough to attempt to improve their PSI (< 3.25). Patients will be seen in clinic at least monthly until treatment is complete and the magnimplant device will be explanted from their sternum.
  Other Names: IDE G090006

SUMMARY:
This study is a Phase 3, multicenter, non-randomized study to evaluate the safety and efficacy of the next-generation outpatient Magnetic Mini-Mover Procedure (3MP) in 15 patients aged 8-14 years for the correction of pectus excavatum ('sunken chest'). 3MP for pectus excavatum uses a magnetically coupled implant to pull the sternum forward and gradually remodel the deformed costal cartilage. The Funding Source for this trial is the FDA Office of Orphan Products Development (Grant #R01 FD003341).

DETAILED DESCRIPTION:
Pectus excavatum is the most common congenital chest wall abnormality in children. The investigators have developed a novel method of achieving gradual deformation/reformation of chest wall cartilage. A magnetic force field is used to apply controlled, sustained force to promote biologic reformation of structural cartilage. A magnet is implanted on the sternum and secured through a 2-inch subxiphoid incision as a one-hour outpatient procedure. The magnet (and sternum) is pulled outward by another magnet suspended in a novel, low-profile, lightweight device previously molded to the patient's anterior chest wall. The low-profile, non-obtrusive anterior chest wall prosthesis is held in place by the force field between the two magnets.

In the single-center, FDA-funded trial (IDE G050196), the investigators tested proof of concept, safety and probable benefit of this procedure in 10. In this Phase III multicenter trial, the investigators will further test the safety and efficacy of the procedure in 15 otherwise healthy patients with moderate-to-severe PE, ages 8 to 14. The investigators will be using the next generation Magnetic Mini-Mover Magnimplant device (IDE G090006), a design the investigators believe is much improved in terms of safety and ease of implantation/explantation. Implantation of the Magnimplant will be accomplished in an outpatient procedure. The investigators will document the rate of correction by comparing chest X-ray measurement of the Pectus Severity Index prior to implantation, to that measured after the magnet is removed. Treatment will last 18-24 months, depending on correction and when the patient has completed his or her pubertal growth spurt, as documented by hand x-ray. Explant of the device will be accomplished in an outpatient procedure. The investigators will document safety with an EKG prior to implantation, one month post-implantation, and finally after the magnet is removed. The investigators will document efficacy by comparing pre- and post-treatment PSI, as well as by evaluating patient satisfaction with a post-procedure Quality of Life-type survey. Long-term follow-up will occur at 6, 12, 18, and 24 months after explantation.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy male or female with pectus excavatum deformity
* Between 8 and 14 years of age (inclusive)
* Pectus Severity Index > 3.5 (normal 2.56). NOTE: A pectus severity index of 3.5 or greater qualifies as a moderate-to-severe deformity, and justifies operative intervention
* Ability to read, speak and understand English
* Onset of rapid growth of puberty documented by hand/wrist x-ray in early to mid-puberty (defined as bone age in females of 7-13 years, and males of 9-14 years)

Exclusion Criteria:

* Other congenital anomalies (including significant skeletal anomalies such as scoliosis, bony fusion involving the cervical vertebrae) not directly related to pectus excavatum
* Bleeding disorders
* Heart disease (including arrhythmia)
* Persons with active implantable medical devices (AIMD) such as pacemakers
* Persons with a relative(s) or close family friend(s) living within their households and having a pacemaker
* Persons with arteriovenous malformations
* Chest deformity more complicated than pectus excavatum (e.g., Poland syndrome)
* Persons for whom a foreign body implant would pose a risk (e.g., immunodeficiency)
* Persons at increased risk for general anesthesia (e.g., history of malignant hyperthermia)
* Respiratory conditions that have required steroid treatment (e.g., prednisone) in the last 3 years
* Pregnancy
* Inability to understand or follow instructions
* Refusal to wear the external brace
* Refusal to undergo monthly chest x-rays
* Inability or refusal to return to UCSF for biweekly follow-up visits for the first month after surgery, and monthly thereafter until explant.
* Inability to obtain pre-approval (authorization) from the patient's insurance carrier

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Harrison, MD, Study Director — University of California, San Francisco; Benjamin Padilla, MD, Principal Investigator — University of California, San Francisco; Lan Vu, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Shriners Hospitals for Children, Sacramento, California
  - UCSF-Benioff Children's Hospital, San Francisco, California
  - Children's Mercy Hospitals, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No
The end results will be published in Journal of Pediatric Surgery June 2017

REFERENCES:
- [Background] Harrison MR, Curran PF, Jamshidi R, Christensen D, Bratton BJ, Fechter R, Hirose S. Magnetic mini-mover procedure for pectus excavatum II: initial findings of a Food and Drug Administration-sponsored trial. J Pediatr Surg. 2010 Jan;45(1):185-91; discussion 191-2. doi: 10.1016/j.jpedsurg.2009.10.032. PMID 20105602
- [Background] Harrison MR, Estefan-Ventura D, Fechter R, Moran AM Jr, Christensen D. Magnetic Mini-Mover Procedure for pectus excavatum: I. Development, design, and simulations for feasibility and safety. J Pediatr Surg. 2007 Jan;42(1):81-5; discussion 85-6. doi: 10.1016/j.jpedsurg.2006.09.042. PMID 17208545
- [Background] Harrison MR, Gonzales KD, Bratton BJ, Christensen D, Curran PF, Fechter R, Hirose S. Magnetic mini-mover procedure for pectus excavatum III: safety and efficacy in a Food and Drug Administration-sponsored clinical trial. J Pediatr Surg. 2012 Jan;47(1):154-9. doi: 10.1016/j.jpedsurg.2011.10.039. PMID 22244409
- See also: Magnetic Mini-Mover Procedure (3MP) Trial — http://pedsurg.ucsf.edu/research/magnetic-mini-mover-trial-study.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: This is a non-randomized study in which otherwise healthy patients, ages 8-14, with severe pectus excavatum (PSI > 3.5) underwent the Magnetic Mini-Mover procedure. The internal magnet, or "Magnimplant" was implanted on the sternum. After surgery and recovery, all subjects were fitted for an orthotic brace, the "Magnatract," which is secured to the patient's chest wall by the attractive force between the coupled internal and external magnets and produces an outward force on the sternum to correct the pectus deformity.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: This is a non-randomized study in which otherwise healthy patients, ages 8-14, with severe pectus excavatum (PSI > 3.5) will undergo the interventional treatment by having outpatient surgery, the Magnetic Mini-Mover procedure, to both place and later explant the experimental Magnimplant or Magnetic Mini-Mover device. After surgery and recovery, all subjects will be fitted for an orthotic brace, which houses the external magnet and records brace-wear compliance. They will undergo 3MP treatment for 24 months. Patients will be seen in clinic at least monthly until treatment is complete.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 12 [8 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Pectus Severity Index (Haller Index) [Mean (Full Range); unit: Ratio] — the Haller Index is calculated as a ratio by measuring across the chest internally from one rib on one side to the rib on the opposite side, then dividing the shortest distance between the spine and sternum.
  Ratio | 4.7 [3.6 to 7.4]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Reactions
Description: All adverse reactions were recorded and reported, including complications from implantation of the device, complications from application of the external device over time (e.g., changes in skin; infection; changes in cardiac electrical function).
Time Frame: During treatment, 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm: All patients who underwent the Magnetic Mini-Mover Procedure
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
Participants
  Discharge home same day | 13
  Normal EKG after implant of magnet | 15
  Surgical site infection | 14
  Intact cables for implant placement | 8

2. Secondary Outcome: Comfort and Brace Wear During Treatment
Description: Comfort of the external brace directly affects compliance (i.e., bracewear) and compliance were be measured throughout treatment. In addition, the satisfaction of the patient and family will be measured using a standard Quality of Life (QOL) questionnaire administered 1 month after implanting the device and 1 month after removing the device.
Time Frame: During treatment, 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
Participants
  Discomfort | 5
  Tolerated Brace wear | 10

3. Secondary Outcome: Chest Wall Correction, by Pectus Severity Index
Description: Though not powered to determine efficacy, preliminary efficacy data, as measured by pre and post treatment Pectus Severity Index (Haller Index), was also collected. Pre-treatment Haller Index was assessed based on computed tomography (CT) of the chest. One month after implant removal, patients underwent repeat chest CT to evaluate chest wall correction.
Time Frame: 24 months
Population: All patients who have received post-treatment chest wall imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 14
Participants
  Improved | 5
  No change | 2
  Worsened | 7
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Other — Pre-treatment and post-treatment Pectus Severity Indices were compared using the Wilcoxon matched-pairs signed rank test; p = 0.486, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Patient Satisfaction During the Treatment
Description: . Patients were asked to fill out questionnaire at 2 intervals: 1 month after explant and 1 year after explant
Time Frame: One month and one year after explant.
Population: 14 Participants offered recommendations at 2 time intervals
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 14
Participants
  Recommend 3MP after 1 month | 11
  Recommend 3MP after 1 year | 11
  Satisfaction with results at 1 month | 9
  Satisfaction with results after 1 year | 8

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Treatment Arm: Magnetic Mini-Mover Procedure (Magnimplant): This is a non-randomized study in which otherwise healthy patients, ages 8-14, with severe pectus excavatum (PSI > 3.5) will undergo the Magnetic Mini-Mover procedure outpatient surgery to both place and later explant the Magnimplant or Magnetic Mini-Mover device. Patients will be required to wear a custom-fitted orthotic brace, which houses the external magnet and records brace-wear compliance. They will undergo 3MP treatment for 24 months.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=15)
Acute cable breakage requiring urgent explant (Product Issues) | 1 — Patient presented to clinic with a sudden anterior movement of the chest and some mild redness of the overlying skin, and a broken cable was discovered on CXR. The implant was removed the following day.
Nonacute cable breakage requiring explant (Cardiac disorders) | 1 — Patient with asymptomatic cable breakage discovered on screening CXR; elected to keep device. Several months later, presented with shortness of breath, symptomatic pericardial effusion, possibly due to device. Device was removed.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=15)
Post-procedure hospitalization for pain control (Surgical and medical procedures) | 1 — Procedure planned as outpatient. However, medical team was unable to adequately control pain in post-operative care unit, and patient was admitted for 3 days for pain control following the procedure.
Wound infection (Skin and subcutaneous tissue disorders) | 1 — Same patient as above (admitted for pain control) developed a superficial surgical site infection 3 weeks after the implant procedure, which resolved with an outpatient course of sulfamethoxazole / trimethoprim.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 — One patient developed a post-operative pneumothorax following the implant procedure and was admitted overnight for chest tube placement and air evacuation.
Rash (Skin and subcutaneous tissue disorders) | 1 — One patient developed a rash on the chest wall from brace wear during warm weather, which resolved with nystatin powder.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less